CLINICAL TRIAL: NCT04077697
Title: Clinical and Prognostic Comparisons Between Invasive Pulmonary Aspergillosis With or Without Invasive Tracheobronchitis During Severe Influenza: a Retrospective Multicenter Cohort Study.
Acronym: ITBA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Lille (Other); Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0047
Record Dates: First submitted 2019-08-21; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Invasive Pulmonary Aspergillosis; Morality
Keywords: invasive pulmonary aspergillosis; Invasive TracheoBronchial Aspergillosis; galactomannan; 1,3-β-D-Glucan; influenza; Intensive Care Unit; mortality
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITBA group: ITBA group is : invasive tracheobronchitis aspergillosis form.
  Interventions: Diagnostic Test: RT-PCR for influenza
- IPA without tracheobronchial involvement: IPA group is : invasive pulmonary aspergillosis without tracheobronchial involvement
  Interventions: Diagnostic Test: RT-PCR for influenza

INTERVENTIONS:
Diagnostic Test: RT-PCR for influenza — influenza real time polymerase chain reaction (RT-PCR) from a nasopharyngeal swab or bronchoalveolar lavage (BAL) fluid.

SUMMARY:
Invasive tracheobronchial aspergillosis (ITBA) is an uncommon, but severe clinical form of Invasive Pulmonary Aspergillosis (IPA) in which the fungal infection is entirely or predominantly confined to the tracheobronchial tree. In view of the limited data concerning critically ill patients admitted to the intensive care unit (ICU) with severe influenza associated with ITBA, the investigators decided to evaluate the differences between the clinical presentations of two invasive infections: ITBA and IPA without tracheobronchial involvement (No ITBA).

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis (IPA) is a well-known complication in severely immunocompromised hosts patients. Recent evidence has identified others populations at risk for IPA, including those with chronic obstructive pulmonary disease (COPD) and advanced cirrhosis patients in intensive care units (ICUs). Moreover, Recently influenza has been identified as a new independent risk factor for IPA and IPA was described as an early complication of influenza. IPA groups different clinical presentations: the classical angio-invasive, the broncho-invasive form and the invasive tracheobronchitis aspergillosis form (ITBA).

ITBA is an infrequent clinical form of IPA with often a fatal outcome, in which Aspergillus infection involves entirely or predominantly the tracheobronchial tree. Early diagnosis of ITBA is based on bronchoscopy examination. Severe influenza is a life-threatening condition where IPA has been repeatedly reported. Little is known on severe influenza infection complicated with IPA and still less with ITBA. Current data on ITBA in critically ill patients hospitalized for severe influenza infection has only been described in single case reports. Because ITBA has been associated with a poorer prognostic than other forms of IPA, this retrospective study aimed to analyze diagnostic and prognostic differences between ITBA and IPA without tracheobronchial lesions, in critically ill patients with influenza infection hospitalized in ICU.

ELIGIBILITY:
Inclusion Criteria:

* all ICU (Intensive care unit) patients
* patients aged from 18 years and more
* All patients hospitalized in ICU with a positive influenza RT-PCR extracted from the registry of the local virology department
* patients with a diagnosis of influenza confirmed by a positive influenza real time polymerase chain reaction (RT-PCR) from nasopharyngeal swab or bronchoalveolar lavage (BAL) fluid, with a concomitant diagnosis of proven or probable/putative IPA and the performing of a bronchoscopy

Exclusion Criteria:

* minor or adult with guardianship
* absence of hospitalization in intensive care
* influenza infection not confirmed by PCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for inclusion were patients with a diagnosis of influenza confirmed by a positive influenza real time polymerase chain reaction (RT-PCR) from nasopharyngeal swab or bronchoalveolar lavage (BAL) fluid, with a concomitant diagnosis of proven or probable/putative IPA and the performing of a bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change of management of ITBA diagnosis criteria | from day 0 to two weeks after the start of the study
  Evolution of the diagnosis criteria of the ITBA

SECONDARY OUTCOMES:
Change of management of ITBA prognosis | from day 0 to two weeks after the start of the study
  Evolution of ITBA prognosis
Change of mortality rate between ITBA group and IPA group | from day 0 to two weeks after the start of the study
  ITBA group is : invasive tracheobronchitis aspergillosis form. IPA group is : invasive pulmonary aspergillosis without tracheobronchial involvement

CONTACTS AND LOCATIONS:
Overall Officials: Elie Zogheib, MD, Principal Investigator — CHU Amiens; Taieb Chouaki, MD, Principal Investigator — CHU Amiens; Hervé Dupont, Pr, Principal Investigator — CHU Amiens; Julien Maizel, Pr, Principal Investigator — CHU Amiens; Rémy Nyga, MD, Principal Investigator — CHU Amiens; Ivona Milic, MD, Principal Investigator — CHU Amiens; Saad NSEIR, Pr, Principal Investigator — CHU Lille; Boualem SENDID, Pr, Principal Investigator — CHU Lille; Malcom LEMYSE, MD, Principal Investigator — CHU Lens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyga R, Maizel J, Nseir S, Chouaki T, Milic I, Roger PA, Van Grunderbeeck N, Lemyze M, Totet A, Castelain S, Slama M, Dupont H, Sendid B, Zogheib E. Invasive Tracheobronchial Aspergillosis in Critically Ill Patients with Severe Influenza. A Clinical Trial. Am J Respir Crit Care Med. 2020 Sep 1;202(5):708-716. doi: 10.1164/rccm.201910-1931OC. PMID 32407157